CLINICAL TRIAL: NCT07146906
Title: An Open-label, Multicenter Study to Assess the Effect of Zigakibart Treatment on Histologic, Circulating, and Excreted Markers of Kidney Disease and Dysfunction in Adult Patients With IgA Nephropathy.
Brief Title: A Study to Assess the Effects of Zigakibart on IgA Nephropathy.
Acronym: SHIFT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFUB523A12201; 2024-519699-24 (Other: EMA (EU CT Number)); U1111-1323-5075 (Other: WHO UTN)
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Immunoglobulin A Nephropathy (IgAN)
Keywords: zigakibart; FUB523; anit-APRIL; SHIFT; IgA nephropathy; IgAN; proteinuria; kidney; biopsy; adults
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a ratio of 1:1 to undergo the on-treatment biopsy at one of two possible timepoints
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- zigakibart (Experimental): zigakibart injections every second week for two years
  Interventions: Biological: zigakibart

INTERVENTIONS:
Biological: zigakibart — zigakibart 600 mg sc injections every second week for 104 weeks (2 years)

SUMMARY:
The purpose of the study is to assess the effect of zigakibart on IgA nephropathy (IgAN) disease progression.

DETAILED DESCRIPTION:
This is an open-label multicenter study where participants are randomized into one of two groups, where the only difference between the groups is the on-treatment biopsy time point, end of the first year of treatment (Group A) or at the end of the second year of treatment (Group B).

The total study duration for each participant may be up to 125 weeks, including the maximum screening period (8 weeks), the treatment period (104 weeks), and the safety follow up period (13 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Primary IgAN, confirmed by kidney biopsy, within 5 years prior to Screening
* eGFR ≥45 mL/min/1.73 m2, based on the 2021 CKD-EPI equation, at Screening
* Persistent proteinuria, defined as either

  * Total Urine Protein ≥0.5 g/day or UPCR ≥0.5 g/g in a 24-hour urine collection, at Screening, despite maximally tolerated dose or poorly tolerated supportive therapy or
  * IgAN diagnosis <6 months prior to Screening with Total Urine Protein >1.5 g/day or UPCR >1.5 g/g in a 24-hour urine collection, at the time of clinical presentation or diagnosis
* Body weight ≥45 kg and body mass index (BMI) ≤35.0 kg/m2, at Screening

Exclusion Criteria:

* Secondary forms of IgAN, as determined by the Investigator, diagnosis of IgA vasculitis, or any other nephropathy or chronic urinary tract disorder
* Total IgG <6.0 g/L at screening
* Any chronic urinary tract disorder, including but not limited to retention, incontinence, and/or recurrent urinary tract infections
* Untreated hypertension or uncontrolled hypertension despite treatment (i.e., resistant hypertension)
* Treatment with complement pathway inhibitors, mycophenolic acids, systemic calcineurin inhibitors or corticosteroids, immunosuppressive or immunomodulatory agents within 12 months prior to screening
* Acute kidney injury (AKI), defined by AKI network criteria, within 4 weeks prior to screening
* Current treatment with anti-APRIL monoclonal antibodies or dual APRIL/BAFF inhibitors or past treatment of the same at any time for >3 consecutive months prior to screening
* Planned initiation of, or recently (within 24 weeks) initiated, treatment with glucagon-like peptide-1 agonists at screening

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2030-07-12 (Estimated); Study Completion 2030-10-18 (Estimated)

PRIMARY OUTCOMES:
Change in mesangial IgA deposition | Baseline to Week 53 or 105
  Change in mesangial IgA deposition as assessed by intensity of immunofluorescence staining

SECONDARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 to Week 118
  Incidence of AEs and SAEs , including changes in vital signs, injection site reactions, laboratory results and Immunoglobulin responses to vaccination qualifying and reported as AEs
Change in MEST-C score | Baseline to Week 53 or 105
  Change in MEST-C, a histologic scoring system used to assess disease prognosis in patients with IgA nephropathy, which includes the components mesangial hypercellularity (M), endocapillary hypercellularity (E), segmental glomerulosclerosis (S), and tubular atrophy/interstitial fibrosis (T), crescents (C).
  All five components are scored by categorical values as listed below, where a higher score indicates involvement or a relatively greater degree of involvement (i.e., more severe pathology).
  1. Mesangial hypercellularity
     * M0 (present in ≤50% of glomeruli)
     * M1 (present in >50% of glomeruli)
  2. Endocapillary hypercellularity
     * E0 (Absent)
     * E1 (Present)
  3. Segmental glomerulosclerosis (more than four mesangial cells)
     * S0 (Absent)
     * S1 (Present)
  4. Tubular atrophy/interstitial fibrosis
     * T0 (0-25% of cortical area)
     * T1 (26-50% of cortical area)
     * T2 (>50% of cortical area)
  5. Cellular or fibrocellular crescents
     * C0 (No crescents)
     * C1 (>25% of glomeruli)
     * C2 (≥25% of glomeruli)
Change in CD68+ cells in glomeruli and tubulo-interstitial compartment | Baseline to Week 53 or 105
  Change in CD68+ cells, which are markers of inflammation
Change in complement component C3c | Baseline to Week 53 or 105
  Change in C3c, which is a marker of complement (part of the immune system) activation
Change in UPCR | Baseline to Week 53 and 105
  Change in the ratio of urine protein to urine creatinine (UPCR), based on 24-hour urine collection
Change in eGFR | Baseline to Week 53 and 105
  Change in estimated glomerular filtration rate (eGFR)
Change in albuminuria | Baseline to Week 53 and 105
  Change in urine albumin - creatinine ratio (UACR), based on 24-hour urine collection
Change in hematuria | Baseline to Week 53 and 105
  Change in presence of red blood cells in urine
Change in serum IgA, IgM and IgG | Baseline to Week 13, 29, 53, 79 and 105
  Immunoglobulin (IgA, IgG and IgM) levels will be assessed from blood samples
Serum zigakibart concentrations | Baseline, Week 13, 29, 66, 79 and 105
  Serum concentration values will be provided
Circulating anti-zigakibart antibodies | Baseline, Week 13, 29, 66, 79 and 105
  Number of participants with circulating binding and neutralizing anti-drug antibodies (ADA/Nab) in blood will be provided

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com